CLINICAL TRIAL: NCT01147627
Title: Comparison of Exenatide, Insulin or Pioglitazone on Glycaemic Control and β-cell Function in Drug-naïve Type 2 Diabetic Patients: A Multicentre Randomized Parallel-group Trial
Brief Title: Effect of Different Interventions on Glycemic Control and β-cell Function in Newly Diagnosed Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Eli Lilly and Company (Industry); Amylin Pharmaceuticals, LLC. (Industry); Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Jianping Weng, professor, vice president, the third affiliated hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-201007-WJP
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2; Newly Diagnosed
Keywords: diabetes mellitus, type 2; newly diagnosed; exenatide; premixed insulin analog; thiazolidinedione; β-cell function; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Commerce; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide (Active Comparator)
  Interventions: Drug: exenatide injection
- Premixed insulin analog (Active Comparator)
  Interventions: Drug: Mixed Protamine Zinc Recombinant Human Insulin Lispro 25R
- pioglitazone (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: exenatide injection — Patients in exenatide group will be treated with exenatide (Byetta®, Eli Lilly and Company) 5 µg BID for the first 4 weeks and then 10 µg BID thereafter.
  Other Names: Byetta®(Eli Lilly and Company)
  Arms: Exenatide
Drug: Mixed Protamine Zinc Recombinant Human Insulin Lispro 25R — Patients in insulin group will be treated with premixed insulin analog (Humalog Mix 25, Eli Lilly and Company). The initial insulin doses are 0.4 IU/kg per day(50% before breakfast and 50% before dinner). Insulin doses are titrated following a forced schedule according to blood glucose before breakfast and dinner.
  Other Names: Humalog Mix 25®（Eli Lilly and Company)
  Arms: Premixed insulin analog
Drug: Pioglitazone — Patients in thiazolidinedione group will be treated with Pioglitazone 30mg daily as single dose. The dose will be increased to 45mg daily after 4 weeks.
  Arms: pioglitazone

SUMMARY:
The purpose of this study is to investigate and evaluate the effects of different interventions (1. exenatide, 2. insulin, 3. thiazolidinedione) on glycemic control and β-cell function in newly diagnosed drug-naïve type 2 diabetic patients.

DETAILED DESCRIPTION:
One of the fundamental defects in type 2 diabetes mellitus is declining β-cell function. Exenatide targets multiple metabolic disturbances in type 2 diabetes and exerts direct effects on β-cell, which indicates that it may not only contribute to the glucose control but also delay disease progression. There are trials demonstrated efficacy, safety and tolerability of exenatide. However, no study has compared the effects of exenatide with other hypoglycemic therapies with β cell protective function in newly diagnosed and drug-naïve type 2 diabetic patients. This current study is thus designed to evaluate the effects of exenatide, insulin and pioglitazone on glycemic control and β-cell function in newly diagnosed drug-naïve type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed type 2 diabetic patients, drug naïve
* age 30~70 years
* HbA1c 7.0~10.0%
* BMI 20~35 kg/m2, stable body weight (≤10% variation) for at least 3 months prior to screening
* female patients of reproductive age should practice a reliable method of birth control throughout the study

Exclusion Criteria:

* acute or severe chronic diabetic complications
* congestive heart failure (NYHA grade Ⅲ~Ⅳ)
* severe gastrointestinal disease
* severe osteoporosis or history of pathological fracture,or use of bisphosphonates preparation
* other severe intercurrent illness
* serum aminotransferase (ALT and AST) level higher than 2 times of the upper normal limits and/or serum creatinie≥133µmol/L (1.5mg/dL)
* tested positive for glutamic acid decarboxylase antibody
* use of weight loss drugs, corticosteroids, drugs known to affect gastrointestinal motility, transplantation medications, or any investigational drug
* history of pancreatitis
* serum triglyceride ≥ 5.0 mmol/L
* pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Weng, Doctor, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (25):
- China (25):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Military General Hospital of Beijing PLA, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Qingyuan People's hospital, Qingyuan, Guangdong
  - The first Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Affiliated hospital of Guangdong medical college, Zhanjiang, Guangdong
  - The first affiliated hospital of Guangxi Medical College, Nanning, Guangxi
  - The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Second Xiangya Hospital of Central-south University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mangolia Medical College, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Zhongda Hospital of Southeast University, Nanjing, Jiangsu
  - China Medical University, Shenyang, Liaoning
  - Xijing Hospital of The Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide: 5 µg was injected twice-daily subcutaneously increasing to 10 µg twice-daily after 4 weeks. Those who experienced hypoglycaemia frequently or could not tolerate adverse events were instructed to reduce the dose to 5 µg twice-daily.
- Premixed Insulin Analog: Premixed insulin was injected twice-daily commencing with 0.4 IU/kg daily, with 50% given 15 minutes before breakfast and dinner respectively
- Pioglitazone: Pioglitazone was commenced at a dose of 30 mg daily, increasing to 45 mg daily after 4 weeks.
Period: Overall Study
Arm/Group | Exenatide | Premixed Insulin Analog | Pioglitazone
Started | 142 | 138 | 136
Completed | 110 | 114 | 118
Not Completed | 32 | 24 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Premixed Insulin Analog | Thiazolidinedione | Total
Number analyzed (Participants) | 142 | 138 | 136 | 416
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 132 | 128 | 129 | 389
  >=65 years | 10 | 10 | 7 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 49.89 (9.64) | 51.39 (9.65) | 49.66 (8.86) | 50.31 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 53 | 150
  Male | 98 | 85 | 83 | 266
Region of Enrollment [Number; unit: participants]
  China | 142 | 138 | 136 | 416

OUTCOME MEASURES:

1. Primary Outcome: the Comparison Between Treatment Groups of the Changes From Baseline in HbA1c at 48 Weeks
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Exenatide | Premixed Insulin Analog | Thiazolidinedione
Number analyzed (Participants) | 110 | 114 | 118
percentage of HbA1c | -1.8 (1.29) | -1.74 (1.16) | -1.47 (1.30)
Statistical Analysis 1: Comparison: Exenatide vs Premixed Insulin Analog vs Thiazolidinedione; Test type: Non-Inferiority or Equivalence — 108 patients in each group was needed to provide 90% power to detect non-inferiority of exenatide, shown by a mean difference of 0.4% in HbA1c change from baseline; p < 0.05, ANCOVA

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <7% and ≤ 6.5% and Effect of Different Interventions on Fasting and Postprandial Plasma Glucose Concentration, Blood Pressure, Lipid Profiles
Time Frame: 48 weeks
Reporting Status: Not Posted

3. Secondary Outcome: β-cell Function (Acute Insulin Response During IVGTT; HOMA-B, Disposition Index and Proinsulin/Insulin Ratio)
Time Frame: 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Safety and Tolerability in Different Groups
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Exenatide | Premixed Insulin Analog | Thiazolidinedione
Serious Adverse Events (participants affected / at risk) | 5/142 | 1/138 | 7/136
Other Adverse Events (participants affected / at risk) | 69/142 | 42/138 | 43/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=142) | Premixed Insulin Analog (N=138) | Thiazolidinedione (N=136)
Cerebral infarction (Vascular disorders) | 1 | 0 | 0
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thigh myofascitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Furuncle and secondary skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Acute nephritis (Renal and urinary disorders) | 0 | 0 | 1
Facial neuritis (Nervous system disorders) | 0 | 0 | 1
Linguinal herniation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cholangiocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Cerebral infarction (Vascular disorders) | 0 | 1 | 0
Cerebral infarction (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=142) | Premixed Insulin Analog (N=138) | Thiazolidinedione (N=136)
Nausea (Gastrointestinal disorders) | 37 | 1 | 1
Vomitting (Gastrointestinal disorders) | 15 | 1 | 1
abdominal pain (Gastrointestinal disorders) | 5 | 2 | 5
diarrhea (Gastrointestinal disorders) | 6 | 1 | 4
abdominal distention (Gastrointestinal disorders) | 8 | 0 | 1
appetite loss (Gastrointestinal disorders) | 8 | 0 | 0
constipation (Gastrointestinal disorders) | 6 | 0 | 1
dizziness (Nervous system disorders) | 18 | 7 | 4
edema (General disorders) | 0 | 0 | 12
numbness (Nervous system disorders) | 4 | 2 | 5
fatigue (General disorders) | 3 | 3 | 4
injection site reaction (Skin and subcutaneous tissue disorders) | 4 | 6 | 0
palpitation (Cardiac disorders) | 4 | 2 | 2
headache (Nervous system disorders) | 3 | 2 | 2
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16 | 13 | 11
blurred vision (Eye disorders) | 2 | 1 | 3
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
chest tightness (Cardiac disorders) | 2 | 0 | 3
rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2
skelalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
toothache (Nervous system disorders) | 3 | 2 | 0
allergy (Immune system disorders) | 0 | 1 | 0
Weight gain (General disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The open-label design, which could have introduced bias by affecting patients' expectations and adherence to therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No